CLINICAL TRIAL: NCT04202861
Title: A Randomised Controlled Trial Evaluating a Novel Individualised Treatment Strategy for Carbapenem-Resistant Gram-Negative Bacteria Infections (iACT)
Brief Title: Evaluating a Novel Individualised Treatment Strategy for Carbapenem-Resistant Gram-Negative Bacteria Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/2880
Record Dates: First submitted 2019-04-14; First posted 2019-12-18 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Antibiotic Therapy

STUDY DESIGN:
Intervention Model Description: The investigators plan to conduct a randomised controlled trial to evaluate a new treatment strategy for CRGNB infections, termed guided antibiotic combination therapy, using the most effective (synergistic and bactericidal) antibiotic combination indicated by iACT. It is an investigator-initiated, two-site, two-arm, open-label, RCT.
  The randomisation will be stratified for the 2 hospitals. At each site, treatments will be randomly assigned to study subjects in a 1:1 ratio using a computer-generated, permuted-block randomisation schedule with a random block size known only to the study biostatistician. Randomisation of participants can be done through a web portal, or through backup randomisation envelopes if internet service is disrupted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in vitro antibiotic combination testing (iACT) (Experimental): For the intervention arm, CRGNB isolates from the index culture should be transported to the Pharmacy Research Lab in Singapore General Hospital as soon as possible to begin iACT. For external sites, a licensed medical courier will be engaged. Once testing is complete, the iACT results will be sent to the physicians and the ID specialist managing the patient. Several antibiotic combinations can usually be used to treat the infection; a subset of results will be published in the iACT report. Participants enrolled into the intervention arm -should ideally be kept on an iACT combination for the required treatment period. However during the treatment period, the treating doctor-in-charge and/or the consulting infectious disease doctor may exercise their discretion in continuing iACT antibiotic combination therapy or modifying the combinations based on their best clinical judgement, according to the clinical conditions and reactions of the patient to the treatment
  Interventions: Diagnostic Test: In vitro antibiotic combination testing (iACT)
- Control (No Intervention): The standard arm will receive standard therapy of either antibiotic monotherapy or unguided combination therapy, a choice based on treating physicians' best clinical judgment. iACT will only be performed on CRGNB isolates from the standard arm at least 30 days after enrolment for collection of microbiological, proteomic and molecular data. Antibiotic combinations found from delayed iACT will be made known to the Infectious Diseases physician caring for the participant.

INTERVENTIONS:
Diagnostic Test: In vitro antibiotic combination testing (iACT) — CRGNB isolates from the index culture will be transported to the Pharmacy Research Lab,SGH for iACT testing. iACT results will be sent to the physicians and ID specialist managing the patient once completed. A subset of results will be published in the iACT report. Participants enrolled into the intervention arm -should ideally be kept on an iACT combination for the required treatment period. However during the treatment period, the treating doctor-in-charge and or the consulting infectious disease doctor may wish to continuing iACT antibiotic combination therapy or modifying the combinations based on their best clinical judgement for the patient.
  Other Names: Intervention Arm
  Arms: in vitro antibiotic combination testing (iACT)

SUMMARY:
Carbapenem-resistant (CR) Gram negative bacteria (GNB) - which are resistant to carbapenems (a last-line potent antibiotic with a high therapeutic index) - are also resistant to all other beta-lactam antibiotics. Most CRGNB are also extensively-drug resistant (XDR) (resistant to all classes of antibiotics except polymyxins and/or tigecycline) or pan-drug resistant (PDR) (resistant to all antibiotics), resulting in a dearth of effective options against these life-threatening infections.

Against CRGNB, standard therapy includes monotherapy (using polymyxins or tigecycline) or unguided antibiotics combination (polymyxins + carbapenem). Unfortunately, CRGNB can develop resistance after antibiotic monotherapy, resulting in the further development of pan-drug resistance. Unguided antibiotic combinations, selected anecdotally based on past experience, are also unlikely to be useful in our local setting, as effective antimicrobial combinations are bacterial-strain specific due to large variation in molecular mechanisms of resistance.Hence, the investigators propose to evaluate the efficacy of a novel treatment strategy using in vitro antibiotic combination testing (iACT) to guide antibiotic combinations in the management of patients with CRGNB infections in a randomised controlled trial (RCT).

DETAILED DESCRIPTION:
The health problem - Antimicrobial resistance (AMR) in GNB and the dearth of therapeutic options AMR, particularly in GNB infections (e.g. Pseudomonas aeruginosa, Enterobacteriaceae and Acinetobacter baumannii), means resistance to multiple or even all available antibiotic classes. The growing incidence of CRGNB and XDRGNB is an urgent global healthcare challenge today. These pathogens are classified as "priority 1" (utmost critical) pathogens by the World Health Organization (WHO). Hsu et al from Singapore has published recently on the estimated prevalence of carbapenem-resistant Enterobacteriaceae (CRE) and carbapenem-resistant A. baumannii (CRA).

Antibiotics are the "foundation" of modern medicine, without which key medical procedures including surgery and chemotherapy for cancer are rendered too dangerous to perform. With the advent of CRGNB, effective antibiotic treatment strategies are now limited. Currently, approximately 700,000 people die from resistant infections every year in the world. It is estimated that by 2050, 10 million lives (1 in 3 The people) per year and a cumulative USD $100 trillion of economic output are at risk due to drug resistant infections, if resistance rates continue to rise unabated. Patel and co-workers observed mortality rates of 40-50% in patients with bloodstream infections caused by CR Klebsiella pneumoniae. Most CRE infections and the transmission of CRE are predominantly linked with healthcare exposure.

Combination therapy - a current mainstay therapeutic option against CRGNB Given the current resistance landscape, coupled with a continued dwindling pipeline of drugs to treat these infections, physicians in Singapore now face a severe lack of effective antimicrobial therapies to treat infections caused by CRGNB. While polymyxin B, an old antibiotic previously forsaken due to an allegedly high rate of toxicities, has been resurrected for such infections, the presence of polymyxin B heteroresistance limits its utility as a monotherapy in severe or deep-seated infections. Currently, antibiotic combination therapy has been adopted by most infectious diseases (ID) physicians locally, as the mainstay treatment against CRGNB infections, because of the theoretical benefits conferred by antibiotic combination therapy (e.g. synergism, prevention of development of resistance). In addition, there is increasing clinical evidence suggesting that antibiotic combination therapy may improve prognosis.

Unfortunately to date, the mortality reduction associated with antibiotic combination therapy in the treatment of CRGNB infections has not been consistently observed across all studies. For example, in a prospective comparison of 55 patients treated for XDR A. baumannii infections, the authors found that the combination of colistin + tigecycline resulted in higher mortality than colistin + a carbapenem when the tigecycline minimum inhibitory concentration (MIC) of the causative pathogen was >2 mg/L (HR = 6.93, 95% CI 1.61-29.78; P= 0.009), suggesting that caution is needed when developing polymyxin combination regimens.

In our local retrospective study, the Investigators have shown that when compared to polymyxins monotherapy or unguided antibiotic combination therapy, the guided selection of a rationally optimised antibiotic combinations was associated with significantly lower rates (by 8 times) of infection-related mortality in patients with XDRGNB infections. In most previous combination therapy studies in the clinical setting, the studies are typically limited by small sample sizes and retrospective nature. To address the ambiguity surrounding the use of polymyxin combinations, three large prospective RCTs are currently underway in Europe and the USA (ClinicalTrials.gov IDs NCT01732250, NCT0159797, NCT03159078)). In these trials, a fixed combination (polymyxins + carbapenem) will be compared to a fixed type of monotherapy (polymyxins alone).

Molecular diversity and complexity in local CRGNB and the implications in antibiotic combination selection Although the aforementioned overseas trials will attempt to address the ambiguity surrounding the use of polymyxin combinations by comparing a fixed combination (colistin + meropenem) to a single monotherapy, the findings of the trials will likely not be generalizable to or applicable in many geographical areas in Asia, especially our local setting, due to the diversity and complexity in the molecular mechanisms of resistance in our local CRGNB strains. Therefore, additional clinical trials will be needed to assess synergy between polymyxins and other agents for specific type pathogens. Such an approach to determining effective antibiotic combinations will be too time-consuming and certainly not cost-effective.

Unlike countries in the United States and Europe, where a predominant K. pneumoniae clonal (ST-258) and resistance type (KPC) is observed, there is greater diversity in Singapore. This greatly complicates management strategies, including the selection of effective combinations for clinical use.

Our local CRE is associated with a variety of resistance mechanisms (e.g. various carbapenemases production in IMPs, KPCs, NDMs, OXA-48, OXA-181, OXA-232, and dual carbapenemases production with/without porin down regulation). The local K. pneumoniae appeared to be of highly varied sequence types (STs) (ST 11, 14, 15, 17, 29, 42, 48, 147, 163, 231, 237, 273, 437, 568, 841, and 885). In addition, the investigators have also detected the presence of mcr-1 novel plasmid that confers resistance to the polymyxins in our CRE isolates that are KPC- or NDM-producers in SGH. For CR A. baumannii, three clones (IC I, IC II, and IC2 II, respectively) from the three outbreaks in 1996, 2001, and 2006 were observed. While these clones harboured carbapenemase producing genes - blaOXA-64, blaOXA-66, and blaOXA-51-like, respectively, blaIMP-4, ISAba1-blaOXA-23-like and blaOXA-58-like have also been described. For CR P. aeruginosa, our local isolates did not belong to any major international clonal complexes such as ST111 and ST235. While carbapenemase production in CR P. aeruginosa is less common, blaIMP and blaVIM have been described. Non-carbapenemase-mediated mechanisms (veb-1 gene +/- efflux pumps +/- porin losses) accounted for carbapenem resistance in local P. aeruginosa strains.

The heterogeneous mechanisms of resistance, coupled with the interplay of multiple resistance mechanisms in local CRGNB, impact on therapy selection decisions and presents as a huge challenge to clinicians locally. The presence of porin mutations and varying levels of porin expression further complicates the pathogen's responses to antibiotic therapy, including combination therapy. For instance, one of the postulated synergy mechanisms is that membrane permeabilisation mediated by polymyxins may enhance the access of carbapenems to their target sites, hence reducing the chances of carbapenem hydrolysis by carbapenemases. This synergistic activity may be diminished in the presence of decreased porin-related permeability, and it is demonstrated that combinations of colistin-doripenem/ertapenem were not synergistic and not bactericidal against isolates with low porin expression. Locally, the investigators have also previously shown that, due to the variability of resistance mechanisms and the interplay between multiple mechanisms, the types of effective antimicrobial combination are bacterial strain-specific. Given the wide variety and permutations of resistance mechanisms, effective antimicrobial combinations are highly varied, and therefore strain-specific testing is required to guide selection of strain-specific combinations in our local setting.

Solving the health problem - Strain-specific combination therapy as a precision therapy against CRGNB In view of the problem described above, the application of "precision medicine" through individualised antimicrobial chemotherapy will be the crux in our combat against CRGNB infections. Strain-specific antibiotics combination testing, in particular, should be performed to guide selection of drugs for combined therapy for the following purposes: Rule out antagonistic antibiotic combinations and ascertain the right and effective antibiotic combination that is synergistic and bactericidal for a specific CRGNB. Currently, in a routine hospital setting, the therapeutic selection for CRGNB is guided by in vitro susceptibility testing (e.g. disk diffusion, Vitek 2), and at best coupled with the determination of MICs (that may require an additional day for results to be available). Currently, this constitutes standard care or best available therapy. However, such traditional single- antibiotic susceptibility results have limited utility in the guiding the selection of combination therapy against CRGNB, as MICs alone are not useful in the prediction of synergistic/bactericidal effect and guide the selection of antibiotics combination therapy, which is required in CRGNB infections where nearly all single antibiotics are ineffective.

In light of the clinical need in our local setting, a prospective in vitro antibiotic combination testing (iACT), with a rapid turn-around time of less than 24 hours (to know an antibiotics combination that is at least inhibitory), was developed to guide physicians in managing patients with CRGNB/XDRGNB infections. The iACT and its workflow were developed at the urgent request of our Infectious Diseases (ID) physicians, after extensive research about the use of iACT for management of patients with CRGNB/XDRGNB infections. Antibiotic combinations, that are shown to be at least inhibitory against the growth of pathogen, will be made known to the requesting ID physician within 18-24 hours. After an additional 20 hours, the bactericidal antibiotics combination will be confirmed with the ID physician. The objective of the iACT is to guide physicians in the selection of an individualised and rationally optimised combination therapy, taking into account the in vitro combination testing results of each strain and the patient's clinical and pharmacokinetic (PK) parameters. To date, the role and feasibility of the iACT, as well as the clinical utility of the service, have been published in a number of retrospective studies. However, iACT is not officially accepted to be used in routine practice in SGH, or anywhere else globally. SGH Translational Medicine Office has recommended that strong evidence with high quality data from prospective, randomised control trials is needed to change current practice.

To fully evaluate the clinical utility of iACT guided therapy, the Investigators propose to conduct an RCT comparing the therapy strategy incorporating iACT to guide selection of antibiotic combinations with current standard therapy. The iACT RCT will overcome the limitations that are inherent in retrospective studies and above-mentioned clinical trials (ClinicalTrials.gov IDs NCT01732250, NCT01597973, NCT03159078) conducted overseas.

Firstly, the RCT design will minimise confounding and allocation bias between treatment arms. Secondly, the use of our novel iACT platform will allow the strain-specific selection of antibiotic combinations against each CRGNB strain in a timely manner, as opposed to using only a single fixed combination in these trials (ClinicalTrials.gov IDs NCT01732250, NCT01597973, NCT03159078). Thirdly, through detailed workup of the presence of various carbapenemases, efflux pumps, and porin loss detection, the Investigators will have detailed description of the molecular mechanisms mediating carbapenem resistance. Such description of the molecular mechanisms will document that our proposed guided therapy strategy is suitable for more than one type of CRGNB infections with variety of resistance mechanisms, and capable of combating against local and global molecular epidemiology of CRGNB infections, strengthening the external validity and applicability of this novel therapy strategy.

Developing new knowledge with scientific and clinical applications Currently, CRGNB are listed as the utmost critical pathogens by the World Health Organization (WHO), for which new and effective treatment strategies against CRGNB is urgently needed. Once completed, our study would represent the first randomised controlled trial that examines the utility of strain-specific antibiotic combination testing in the treatment of CRGNB infections. If our hypothesis is proven, this guided therapy strategy can change current practice paradigms in the treatment of CRGNB both locally and internationally, and provide a novel solution to the management of CRGNB infections. Given the heterogeneity of patients with CRGNB infections, our proposed RCT unequivocally addresses the challenges in treating CRGNB infection in ways that is otherwise not possible (e.g. ClinicalTrials.gov IDs NCT01732250, NCT01597973, NCT03159078). Through the description of the molecular epidemiology of CRGNB infections in our study, the Investigators will provide new insight into the complicated resistance mechanisms common in our local CRGNB strains. The investigators anticipate that the findings of this study will drive further research, particularly translational research, to further enrich knowledge, and improve management, of CRGNB infections.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient at the time of enrolment.
2. Age ≥16 years.
3. An ongoing infection as defined by the published Centers for Disease Control and Prevention (CDC) /National Healthcare Safety Network (NHSN) or Infectious Diseases Society of America (IDSA) guidelines; Section 16.1-16.6 Appendix specifies the most common examples expected in this study.
4. Positive culture of CRGNB isolates from relevant clinical sites (i.e. samples that are not obtained for surveillance purposes, such as rectal swabs)
5. No more than 5 calendar days has elapsed since the first positive culture collection.

Exclusion Criteria:

1. Unable to provide consent AND have no legal representative (LR).
2. Subjects on palliative care or with less than 24 hours of life expectancy (as discussed with their primary physicians).
3. Colonisation only, which is defined as positive isolation of CRGNB isolated at screening sites (e.g., rectal swabs) only
4. Prior recruitment into this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
30-day all cause mortality rate post therapy initiation after randomization | 30 days
  We define this as all cause mortality as death of any cause. We aim to compare the difference in 30-day all cause mortality rates post therapy initiation between both arms

SECONDARY OUTCOMES:
30-day infection-related mortality post therapy initiation after randomization | 30 days
  We defined infectious disease-related mortality as death that could be attributed to infectious disease as either the immediate or underlying cause. The term "immediate cause of death" is defined as the infectious disease directly leading to death, and the term "underlying cause of death" is defined as the infectious disease initiated the sequence of events that led directly to death. The Infectious Diseases physicians of the recruited subjects will decide if the mortality at 30 days is infection-related
Microbiological clearance | Day 7 post randomisation
  We defined microbiological clearance as observation of microbiological eradication of the intended pathogen at the original site of isolation

CONTACTS AND LOCATIONS:
Overall Officials: Andrea LH Kwa, PharmD, Principal Investigator — Singapore General Hospital
Locations (1):
- Andrea Lay Hoon KWA (SGH), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai Y, Chua NG, Lim TP, Teo JQ, Lee W, Kurup A, Koh TH, Tan TT, Kwa AL. From Bench-Top to Bedside: A Prospective In Vitro Antibiotic Combination Testing (iACT) Service to Guide the Selection of Rationally Optimized Antimicrobial Combinations against Extensively Drug Resistant (XDR) Gram Negative Bacteria (GNB). PLoS One. 2016 Jul 21;11(7):e0158740. doi: 10.1371/journal.pone.0158740. eCollection 2016. PMID 27441603
- [Background] Cai Y, Lim TP, Teo J, Sasikala S, Lee W, Hong Y, Chan EC, Tan TY, Tan TT, Koh TH, Hsu LY, Kwa AL. In Vitro Activity of Polymyxin B in Combination with Various Antibiotics against Extensively Drug-Resistant Enterobacter cloacae with Decreased Susceptibility to Polymyxin B. Antimicrob Agents Chemother. 2016 Aug 22;60(9):5238-46. doi: 10.1128/AAC.00270-16. Print 2016 Sep. PMID 27324776
- [Background] Cai B, Cai Y, Liew YX, Chua NG, Teo JQ, Lim TP, Kurup A, Ee PL, Tan TT, Lee W, Kwa AL. Clinical Efficacy of Polymyxin Monotherapy versus Nonvalidated Polymyxin Combination Therapy versus Validated Polymyxin Combination Therapy in Extensively Drug-Resistant Gram-Negative Bacillus Infections. Antimicrob Agents Chemother. 2016 Jun 20;60(7):4013-22. doi: 10.1128/AAC.03064-15. Print 2016 Jul. PMID 27090177
- [Background] Lim TP, Tan TY, Lee W, Sasikala S, Tan TT, Hsu LY, Kwa AL. In-vitro activity of polymyxin B, rifampicin, tigecycline alone and in combination against carbapenem-resistant Acinetobacter baumannii in Singapore. PLoS One. 2011 Apr 21;6(4):e18485. doi: 10.1371/journal.pone.0018485. PMID 21533030
- [Background] Lim TP, Lee W, Tan TY, Sasikala S, Teo J, Hsu LY, Tan TT, Syahidah N, Kwa AL. Effective antibiotics in combination against extreme drug-resistant Pseudomonas aeruginosa with decreased susceptibility to polymyxin B. PLoS One. 2011;6(12):e28177. doi: 10.1371/journal.pone.0028177. Epub 2011 Dec 5. PMID 22162759
- [Background] Lim TP, Cai Y, Hong Y, Chan EC, Suranthran S, Teo JQ, Lee WH, Tan TY, Hsu LY, Koh TH, Tan TT, Kwa AL. In vitro pharmacodynamics of various antibiotics in combination against extensively drug-resistant Klebsiella pneumoniae. Antimicrob Agents Chemother. 2015 May;59(5):2515-24. doi: 10.1128/AAC.03639-14. Epub 2015 Feb 17. PMID 25691628
- [Background] Hsu LY, Apisarnthanarak A, Khan E, Suwantarat N, Ghafur A, Tambyah PA. Carbapenem-Resistant Acinetobacter baumannii and Enterobacteriaceae in South and Southeast Asia. Clin Microbiol Rev. 2017 Jan;30(1):1-22. doi: 10.1128/CMR.masthead.30-1. Epub 2016 Oct 19. PMID 27795305
- [Background] Patel G, Huprikar S, Factor SH, Jenkins SG, Calfee DP. Outcomes of carbapenem-resistant Klebsiella pneumoniae infection and the impact of antimicrobial and adjunctive therapies. Infect Control Hosp Epidemiol. 2008 Dec;29(12):1099-106. doi: 10.1086/592412. PMID 18973455
- [Background] Perez F, Endimiani A, Ray AJ, Decker BK, Wallace CJ, Hujer KM, Ecker DJ, Adams MD, Toltzis P, Dul MJ, Windau A, Bajaksouzian S, Jacobs MR, Salata RA, Bonomo RA. Carbapenem-resistant Acinetobacter baumannii and Klebsiella pneumoniae across a hospital system: impact of post-acute care facilities on dissemination. J Antimicrob Chemother. 2010 Aug;65(8):1807-18. doi: 10.1093/jac/dkq191. Epub 2010 May 31. PMID 20513702
- [Background] Perez F, Van Duin D. Carbapenem-resistant Enterobacteriaceae: a menace to our most vulnerable patients. Cleve Clin J Med. 2013 Apr;80(4):225-33. doi: 10.3949/ccjm.80a.12182. PMID 23547093
- [Background] Cai Y, Lee W, Kwa AL. Polymyxin B versus colistin: an update. Expert Rev Anti Infect Ther. 2015;13(12):1481-97. doi: 10.1586/14787210.2015.1093933. Epub 2015 Oct 21. PMID 26488563
- [Background] Li J, Rayner CR, Nation RL, Owen RJ, Spelman D, Tan KE, Liolios L. Heteroresistance to colistin in multidrug-resistant Acinetobacter baumannii. Antimicrob Agents Chemother. 2006 Sep;50(9):2946-50. doi: 10.1128/AAC.00103-06. PMID 16940086
- [Background] Falagas ME, Lourida P, Poulikakos P, Rafailidis PI, Tansarli GS. Antibiotic treatment of infections due to carbapenem-resistant Enterobacteriaceae: systematic evaluation of the available evidence. Antimicrob Agents Chemother. 2014;58(2):654-63. doi: 10.1128/AAC.01222-13. Epub 2013 Sep 30. PMID 24080646
- [Background] Qureshi ZA, Paterson DL, Potoski BA, Kilayko MC, Sandovsky G, Sordillo E, Polsky B, Adams-Haduch JM, Doi Y. Treatment outcome of bacteremia due to KPC-producing Klebsiella pneumoniae: superiority of combination antimicrobial regimens. Antimicrob Agents Chemother. 2012 Apr;56(4):2108-13. doi: 10.1128/AAC.06268-11. Epub 2012 Jan 17. PMID 22252816
- [Background] Daikos GL, Tsaousi S, Tzouvelekis LS, Anyfantis I, Psichogiou M, Argyropoulou A, Stefanou I, Sypsa V, Miriagou V, Nepka M, Georgiadou S, Markogiannakis A, Goukos D, Skoutelis A. Carbapenemase-producing Klebsiella pneumoniae bloodstream infections: lowering mortality by antibiotic combination schemes and the role of carbapenems. Antimicrob Agents Chemother. 2014;58(4):2322-8. doi: 10.1128/AAC.02166-13. Epub 2014 Feb 10. PMID 24514083
- [Background] Rigatto MH, Vieira FJ, Antochevis LC, Behle TF, Lopes NT, Zavascki AP. Polymyxin B in Combination with Antimicrobials Lacking In Vitro Activity versus Polymyxin B in Monotherapy in Critically Ill Patients with Acinetobacter baumannii or Pseudomonas aeruginosa Infections. Antimicrob Agents Chemother. 2015 Oct;59(10):6575-80. doi: 10.1128/AAC.00494-15. Epub 2015 Aug 10. PMID 26259799
- [Background] Petrosillo N, Giannella M, Antonelli M, Antonini M, Barsic B, Belancic L, Inkaya A C, De Pascale G, Grilli E, Tumbarello M, Akova M. Clinical experience of colistin-glycopeptide combination in critically ill patients infected with Gram-negative bacteria. Antimicrob Agents Chemother. 2014;58(2):851-8. doi: 10.1128/AAC.00871-13. Epub 2013 Nov 25. PMID 24277037
- [Background] Sirijatuphat R, Thamlikitkul V. Preliminary study of colistin versus colistin plus fosfomycin for treatment of carbapenem-resistant Acinetobacter baumannii infections. Antimicrob Agents Chemother. 2014 Sep;58(9):5598-601. doi: 10.1128/AAC.02435-13. Epub 2014 Jun 30. PMID 24982065
- [Background] Chen Z, Chen Y, Fang Y, Wang X, Chen Y, Qi Q, Huang F, Xiao X. Meta-analysis of colistin for the treatment of Acinetobacter baumannii infection. Sci Rep. 2015 Nov 24;5:17091. doi: 10.1038/srep17091. PMID 26597507
- [Background] Pogue JM, Kaye KS. Is there really no benefit to combination therapy with colistin? Expert Rev Anti Infect Ther. 2013 Sep;11(9):881-4. doi: 10.1586/14787210.2013.827881. PMID 24053270
- [Background] Cheng A, Chuang YC, Sun HY, Sheng WH, Yang CJ, Liao CH, Hsueh PR, Yang JL, Shen NJ, Wang JT, Hung CC, Chen YC, Chang SC. Excess Mortality Associated With Colistin-Tigecycline Compared With Colistin-Carbapenem Combination Therapy for Extensively Drug-Resistant Acinetobacter baumannii Bacteremia: A Multicenter Prospective Observational Study. Crit Care Med. 2015 Jun;43(6):1194-204. doi: 10.1097/CCM.0000000000000933. PMID 25793437
- [Background] Teo JQ, Cai Y, Lim TP, Tan TT, Kwa AL. Carbapenem Resistance in Gram-Negative Bacteria: The Not-So-Little Problem in the Little Red Dot. Microorganisms. 2016 Feb 16;4(1):13. doi: 10.3390/microorganisms4010013. PMID 27681907
- [Background] Teo JWP, La MV, Krishnan P, Ang B, Jureen R, Lin RTP. Enterobacter cloacae producing an uncommon class A carbapenemase, IMI-1, from Singapore. J Med Microbiol. 2013 Jul;62(Pt 7):1086-1088. doi: 10.1099/jmm.0.053363-0. Epub 2013 Apr 4. PMID 23558141
- [Background] Koh TH, Babini GS, Woodford N, Sng LH, Hall LM, Livermore DM. Carbapenem-hydrolysing IMP-1 beta-lactamase in Klebsiella pneumoniae from Singapore. Lancet. 1999 Jun 19;353(9170):2162. doi: 10.1016/s0140-6736(05)75604-x. No abstract available. PMID 10382730
- [Background] Koh TH, Sng LH, Babini GS, Woodford N, Livermore DM, Hall LM. Carbapenem-resistant Klebsiella pnuemoniae in Singapore producing IMP-1 beta-lactamase and lacking an outer membrane protein. Antimicrob Agents Chemother. 2001 Jun;45(6):1939-40. doi: 10.1128/AAC.45.6.1939-1940.2001. No abstract available. PMID 11407332
- [Background] Koh TH, Cao D, Shan QY, Bacon A, Hsu LY, Ooi EE. Acquired carbapenemases in Enterobactericeae in Singapore, 1996-2012. Pathology. 2013 Oct;45(6):600-3. doi: 10.1097/PAT.0b013e3283650b1e. PMID 24018814
- [Background] Balm MN, La MV, Krishnan P, Jureen R, Lin RT, Teo JW. Emergence of Klebsiella pneumoniae co-producing NDM-type and OXA-181 carbapenemases. Clin Microbiol Infect. 2013 Sep;19(9):E421-3. doi: 10.1111/1469-0691.12247. Epub 2013 May 13. PMID 23668475
- [Background] Balm MN, Ngan G, Jureen R, Lin RT, Teo J. Molecular characterization of newly emerged blaKPC-2-producing Klebsiella pneumoniae in Singapore. J Clin Microbiol. 2012 Feb;50(2):475-6. doi: 10.1128/JCM.05914-11. Epub 2011 Nov 23. PMID 22116160
- [Background] Teo J, Ngan G, Balm M, Jureen R, Krishnan P, Lin R. Molecular characterization of NDM-1 producing Enterobacteriaceae isolates in Singapore hospitals. Western Pac Surveill Response J. 2012 Mar 29;3(1):19-24. doi: 10.5365/WPSAR.2011.2.4.010. Print 2012 Jan. PMID 23908903
- [Background] Teo JQ, Ong RT, Xia E, Koh TH, Khor CC, Lee SJ, Lim TP, Kwa AL. mcr-1 in Multidrug-Resistant blaKPC-2-Producing Clinical Enterobacteriaceae Isolates in Singapore. Antimicrob Agents Chemother. 2016 Sep 23;60(10):6435-7. doi: 10.1128/AAC.00804-16. Print 2016 Oct. No abstract available. PMID 27503652
- [Background] Hawkey PM. Multidrug-resistant Gram-negative bacteria: a product of globalization. J Hosp Infect. 2015 Apr;89(4):241-7. doi: 10.1016/j.jhin.2015.01.008. Epub 2015 Feb 4. PMID 25737092
- [Background] Hong JH, Clancy CJ, Cheng S, Shields RK, Chen L, Doi Y, Zhao Y, Perlin DS, Kreiswirth BN, Nguyen MH. Characterization of porin expression in Klebsiella pneumoniae Carbapenemase (KPC)-producing K. pneumoniae identifies isolates most susceptible to the combination of colistin and carbapenems. Antimicrob Agents Chemother. 2013 May;57(5):2147-53. doi: 10.1128/AAC.02411-12. Epub 2013 Mar 4. PMID 23459476
- [Background] Shields RK, Nguyen MH, Potoski BA, Press EG, Chen L, Kreiswirth BN, Clarke LG, Eschenauer GA, Clancy CJ. Doripenem MICs and ompK36 porin genotypes of sequence type 258, KPC-producing Klebsiella pneumoniae may predict responses to carbapenem-colistin combination therapy among patients with bacteremia. Antimicrob Agents Chemother. 2015 Mar;59(3):1797-801. doi: 10.1128/AAC.03894-14. Epub 2014 Dec 22. PMID 25534733
- [Background] Clancy CJ, Chen L, Hong JH, Cheng S, Hao B, Shields RK, Farrell AN, Doi Y, Zhao Y, Perlin DS, Kreiswirth BN, Nguyen MH. Mutations of the ompK36 porin gene and promoter impact responses of sequence type 258, KPC-2-producing Klebsiella pneumoniae strains to doripenem and doripenem-colistin. Antimicrob Agents Chemother. 2013 Nov;57(11):5258-65. doi: 10.1128/AAC.01069-13. Epub 2013 Aug 12. PMID 23939888